CLINICAL TRIAL: NCT01275794
Title: Screening Epidemiological Program on Compensation Evaluation of DM Type 2 Patients on OAD Monotherapy and Physicians Satisfaction of Their Usage
Brief Title: Screening Epidemiological Program on Compensation Evaluation of Diabetes Mellitus Type 2 (DMT2) Patients on Oral Anti-diabetic (OAD) Monotherapy and Physicians Satisfaction of Their Usage
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-ONG-2010/1
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients have an established diagnosis of T2D, Age 35 years and more, Experience of therapy with one OAD during the from 6 months to 5 years before the registration in the Program

SUMMARY:
The purpose of the study is assessment of glycemic control and physicians satisfaction with results of DM2 OAD monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients have an established diagnosis of T2D
* Experience of therapy with one OAD during the from 6 months to 5 years before the registration in the Program

Exclusion Criteria:

* Experience of therapy with two or more OADs and/or insulin therapy and/or incretin mimetics (exenatide) at any time before registration in the Program
* Absence of changes in HbAc1 level during the last year before registration in the Program

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1849 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess levels of compensation of T2D by HbA1c levels in patients on OAD monotherapy | 1 visit within 4 month
To assess frequency of target levels of HbA1c ≤ 7% in patients with T2D during OAD monotherapy | 1 visit within 4 month

SECONDARY OUTCOMES:
To assess fasting glycemia in patients with T2D on OAD monotherapy | 1 visit within 4 month
To assess postprandial levels of glycemia in patients with T2D during OAD monotherapy | 1 visit within 4 month
To evaluate the physicians' satisfaction with the results of OAD monotherapy in patients with Typ 2 Diabetes (T2D) | 1 visit within 4 month
To compare the results of OAD monotherapy in different groups of patients | 1 visit within 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Study Director — AstraZeneca
Locations (23):
- Russia (23):
  - Research Site, Arkhangelsk
  - Research Site, Astrakhan
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Khemerovo
  - Research Site, Kirov
  - Research Site, Kurgan
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Perm
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Samara
  - Research Site, Seversk
  - Research Site, Smolensk
  - Research Site, St-Peterburg
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Yaroslavl
  - Research Site, Yoshkar-Ola